CLINICAL TRIAL: NCT06574646
Title: Visual Acuity Outcome Differences Between the Alcon Vivity Toric IOL and RxSight LAL+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Associates (Other)
Responsible Party: Principal Investigator, Cathleen McCabe MD, Medical Director, The Eye Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A126-101
Record Dates: First submitted 2024-08-09; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cataract
Keywords: intraocular lens; LAL+; Clareon Vivity Toric IOLs
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LAL+ (Experimental)
  Interventions: Device: LAL+
- Clareon Vivity Toric IOLs (Active Comparator)
  Interventions: Device: Clareon Vivity Toric IOL

INTERVENTIONS:
Device: LAL+ — LAL+ IOL allows for refractive error (both sphere and cylinder) enhancements post-IOL implantation by exposing the IOL to ultraviolet (UV) light through a series of noninvasive treatments with a Light Delivery Device.
  Arms: LAL+
Device: Clareon Vivity Toric IOL — Clareon Vivity Toric IOL utilizes an extended depth of focus (EDOF) design, which incorporates nondiffractive wavefront shaping (X-WAVE) technology.
  Arms: Clareon Vivity Toric IOLs

SUMMARY:
Phase 1 will be ambispective, multi-site, single arm study in age-related cataract patients with regular astigmatism, who were bilaterally treated with the LAL+ IOLs

Phase 2 will be a prospective, randomized, unmasked, comparative, multi-site study with 90 days of follow up. Subjects will be randomized in a 1:1 manner to LAL+ or Clareon VIvity Toric IOLs.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥45) subjects who are astigmatic and require bilateral, routine small-incision, surgery for age-related cataracts with femtosecond laser;
* All subjects will be required to be targeted for refractive emmetropia (plano or first minus closest to plano);
* Subjects will have an expected monocular BCDVA outcomes of 20/25 or better in the opinion of the investigator;
* Subjects will have regular corneal astigmatism (1.00 to 2.00 D), which can be corrected with a toric power IOL of T3-T5;
* Subjects will be required to have a dilated pupil diameter of 7 mm or greater in both eyes;

Exclusion Criteria:

* Moderate-severe corneal pathology;

  * Irregular astigmatism;
  * Subject desire monovision correction;
  * Preexisting macular disease or other retinal degenerative diseases that is expected to cause future vision loss;
  * History of glaucoma;
  * Severe dry eye disease;
  * History of uveitis;
  * History of ocular herpes simplex virus;
  * History of nystagmus;
  * Zonular laxity or dehiscence;
  * History psueudoexfoliation;
  * History of corneal refractive and intraocular surgery or requiring any other planned ocular surgical procedures;
  * Currently taking systemic medication that may increase sensitivity to UV light or that may cause toxicity to the retina;
  * Pregnant or breastfeeding.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Binocular photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 cm | at the 90-day post-op visit or at least 1 week after final lock-in if longer than 3 months for LAL+ implanted subjects and >2 weeks post YAG, if done.
  Binocular photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 cm

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen M McCabe, MD, Principal Investigator — The Eye Associates of Manatee
Locations (1):
- The Eye Associates of Manatee, LLP, Bradenton, Florida, United States